CLINICAL TRIAL: NCT06664580
Title: Enhancing Nutritional Health and Patient Satisfaction Five Years After Metabolic Bariatric Surgery with Targeted Supplementation
Brief Title: Nutritional Health and Satisfaction After Bariatric Surgery: a Five-Year Retrospective Study
Status: Completed | Type: Observational
Sponsor: San Raffaele Telematic University (Other)
Responsible Party: Principal Investigator, Mauro Lombardo, Associate Professor of Nutrition Sciences, University of Rome Tor Vergata
Other Study IDs: 100/SR/24
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Obesity and Overweight; Nutritional Deficiency; Bariatric Surgery
Keywords: Metabolic Bariatric Surgery; Laparoscopic Sleeve Gastrectomy; Roux-en-Y Gastric Bypass; Excess Weight Loss; Iron Deficiency; Vitamin D Deficiency; Quality of Life Post-Surgery; Targeted Supplementation
MeSH Terms: conditions — Obesity; Overweight; Malnutrition; Iron Deficiencies; Vitamin D Deficiency | interventions — Bariatric Surgery; Weights and Measures; Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post-Metabolic Bariatric Surgery Patients: A cohort of 249 patients who underwent metabolic bariatric surgery, including various procedures such as Laparoscopic Sleeve Gastrectomy (LSG) and Roux-en-Y Gastric Bypass (RYGB), with follow-up on long-term outcomes related to weight maintenance, nutritional deficiencies, and patient satisfaction
  Interventions: Other: Metabolic Bariatric Surgery Procedures

INTERVENTIONS:
Other: Metabolic Bariatric Surgery Procedures — Observational analysis of various metabolic bariatric surgeries, including LSG, RYGB, and OAGB, focusing on long-term outcomes related to weight maintenance, nutritional health, and patient satisfaction.
  Other Names: weight; bariatric; nutrition

SUMMARY:
A retrospective study analyzing long-term outcomes of metabolic bariatric surgery (MBS) with a focus on weight loss, nutritional deficiencies, and patient satisfaction over a five-year follow-up. This study evaluates outcomes for different surgical procedures, including Laparoscopic Sleeve Gastrectomy (LSG), Roux-en-Y Gastric Bypass (RYGB), and other MBS techniques. The findings aim to provide insight into optimal nutritional management and patient care following bariatric surgery.

DETAILED DESCRIPTION:
This study retrospectively examines 249 patients who underwent metabolic bariatric surgery at a specialized center between 2012 and 2017. It evaluates long-term outcomes including weight loss, excess weight loss percentage (%EWL), and nutritional deficiencies, with a specific focus on the effectiveness of targeted supplementation protocols to improve nutritional health post-surgery. The study analyzes different surgical procedures, including LSG, RYGB, and others, comparing primary and revision surgeries. Nutritional deficiencies in essential vitamins and minerals are assessed, highlighting the need for individualized supplementation based on the type of surgery and patient adherence.

Key objectives include:

1. Assessing long-term weight loss and maintenance across different MBS procedures.
2. Identifying the prevalence of nutritional deficiencies, particularly for iron, vitamin D, and B12.
3. Evaluating patient satisfaction and quality of life improvements following MBS.

Data were collected from electronic clinical records and include anthropometric data, biochemical markers, and self-reported supplement use. Findings emphasize the importance of targeted supplementation and regular monitoring to address persistent deficiencies. The study contributes to understanding optimal long-term care strategies for MBS patients and underscores the importance of personalized nutritional support post-surgery.

ELIGIBILITY:
Inclusion criteria: Patients aged 18 to 65 years who underwent metabolic bariatric surgery (MBS) at the Specialized Bariatric Center between 2012 and 2017, with a follow-up period of at least five years post-surgery.

Exclusion criteria: Individuals with a history of alcoholism, severe social anxiety impacting post-operative care participation, recent neoplastic disease diagnoses, neurocognitive disorders, or other systemic diseases potentially affecting quality of life and long-term outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults who underwent metabolic bariatric surgery, including LSG and RYGB, at a specialized center, with a focus on long-term outcomes in weight maintenance, nutritional health, and patient satisfaction
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Excess Weight Loss (%EWL) | The percentage of excess weight lost relative to baseline, calculated to assess long-term weight maintenance following different metabolic bariatric surgeries.
  5 years post-surgery

SECONDARY OUTCOMES:
Incidence of Nutritional Deficiencies | 5 years post-surgery
  Rate of nutritional deficiencies, specifically in iron, vitamin D, and vitamin B12, following metabolic bariatric surgery, with a focus on patients receiving targeted supplementation.
Patient Satisfaction and Quality of Life | 5 years post-surgery
  Self-reported patient satisfaction and quality of life improvement post-surgery, assessed through a custom survey.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and the retrospective nature of the study, which limits consent for data sharing beyond the initial research purposes. Aggregated study results and relevant findings are available upon reasonable request.

REFERENCES:
- [Background] Heusschen L, Berendsen AAM, Deden LN, Hazebroek EJ, Aarts EO. Nutritional Deficiencies 3 Years After Sleeve Gastrectomy Can Be Limited by a Specialized Multivitamin Supplement. Obes Surg. 2022 Nov;32(11):3561-3570. doi: 10.1007/s11695-022-06256-w. Epub 2022 Aug 26. PMID 36018421
- [Background] Noria SF, Shelby RD, Atkins KD, Nguyen NT, Gadde KM. Weight Regain After Bariatric Surgery: Scope of the Problem, Causes, Prevention, and Treatment. Curr Diab Rep. 2023 Mar;23(3):31-42. doi: 10.1007/s11892-023-01498-z. Epub 2023 Feb 8. PMID 36752995
- [Derived] Gorini S, Camajani E, Franchi A, Cava E, Gentileschi P, Bellia A, Karav S, Sbraccia P, Caprio M, Lombardo M. Enhancing nutritional health and patient satisfaction five years after metabolic bariatric surgery with targeted supplementation. J Transl Med. 2025 Feb 21;23(1):216. doi: 10.1186/s12967-025-06224-9. PMID 39984967
- See also: Collaboration Agreement on: 'RETROSPECTIVE ASSESSMENT OF WEIGHT LOSS AND NUTRITIONAL DEFICIENCIES IN PATIENTS UNDERGOING BARIATRIC SURGERY' Between: Nutrition Unit, San Raffaele Telematic University (hereafter 'Unit'), e UOC Internal Medicine — https://drive.google.com/drive/u/0/folders/14aOTiUJ0qTP_hVzt0Nl2w3hQRqE18MnK